CLINICAL TRIAL: NCT05126238
Title: A Lithium-Based Medication to Improve Neurological Outcomes After Surgical Carotid Reconstruction: A Double-Blind, Placebo Control Randomized Trial (BINOS)
Brief Title: A Lithium-Based Medication to Improve Neurological Outcomes After Surgical Carotid Reconstruction
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Decision of the local ethics committee
Sponsor: Negovsky Reanimatology Research Institute (Other Government)
Collaborators: Demikhov Municipal Clinical Hospital 68 (Other Government)
Responsible Party: Principal Investigator, Valery Likhvantsev, MD, Head of the Research V. Negovsky Reanimatology Research Institute, Negovsky Reanimatology Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BINOS
Record Dates: First submitted 2021-10-01; First posted 2021-11-18 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Carotid Artery Diseases; Carotid Artery Stenosis
Keywords: Carotid artery diseases; Carotid artery stenosis; Carotid artery surgery; Lithium; Neurocognitive disorders; Postoperative cognitive disorders; Postoperative delirium; Emergence delirium; Agitation; Stroke; Neuroinflammation
MeSH Terms: conditions — Carotid Artery Diseases; Carotid Stenosis; Neurocognitive Disorders; Postoperative Cognitive Complications; Emergence Delirium; Psychomotor Agitation; Stroke; Neuroinflammatory Diseases | interventions — Lithium Carbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lithium (Experimental): In preoperative period patients will take 300mg of lithium carbonate on 1-1-1 regimen during 2 days prior to surgery. On the day of surgery, they will take 300mg of lithium carbonate 2 hours before surgery. After the surgery, patients will take 300mg of lithium carbonate in the afternoon and 300mg of lithium carbonate in the evening.
  Interventions: Drug: Lithium Carbonate
- Placebo (Placebo Comparator): In preoperative period patients will take placebo on 1-1-1 regimen during 2 days prior to surgery. On the day of surgery, they will take placebo 2 hours before surgery. After the surgery, patients will take placebo in the afternoon and in the evening.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lithium Carbonate — In preoperative period patients will take 300 mg of lithium carbonate on 1-1-1 regimen during 2 days prior to surgery. On the day of surgery they will take 300mg of lithium carbonate 2 hours before surgery.
  Arms: Lithium
Drug: Placebo — In preoperative period patients will take placebo on 1-1-1 regimen during 2 days prior to surgery. On the day of surgery they will placebo 2 hours before surgery.
  Arms: Placebo

SUMMARY:
There are 10.3 million cases of stroke registered in the world every year; 63% of them lead to death. According to World Health Organization, stroke is one of the most important risk factors of death and early disability.

Carotid artery surgery is a gold standard of hemodynamically significant carotid artery disease treatment. According to some trials, carotid artery surgery decreases the 2-years mortality.

The most important part of carotid artery surgery is a temporary absence of blood flow in the carotid artery. The duration of this period is a crucial characteristic of this type of surgery. The absence of blood flow leads to brain ischemia which is the risk factor of postoperative neurocognitive disorders such as emergence delirium, postoperative delirium and postoperative cognitive dysfunction.

Some surgical and non-surgical methods for brain protection were evaluated. According to recent data, there is no evidence of effective pharmacological protective methods that can decrease brain damage during carotid artery surgery.

Nevertheless, some trials demonstrated that using lithium-based medications for patients with a stroke can reduce the volume of the stroke. Therefore, the investigators want to check the hypothesis that using lithium-based medication in the preoperative period can reduce brain damage during carotid artery surgery.

The objectives of this trial:

1. To determine if Lithium carbonate is superior to placebo for the occurrence of emergence delirium, agitation, postoperative delirium and postoperative cognitive dysfunction.
2. To determine if Lithium carbonate is non-inferior to placebo for the occurrence of a new arrhythmia, leukocytosis, acute kidney injury, seizure disorders, diarrhea, nausea, and vomit.

DETAILED DESCRIPTION:
There are 10.3 million cases of stroke registered in the world every year; 63% of them lead to death. According to World Health Organization, stroke is one of the most important risk factors of death and early disability.

Carotid artery surgery is a gold standard of hemodynamically significant carotid artery disease treatment. According to some trials, carotid artery surgery decreases the 2-years mortality.

The most important part of carotid artery surgery is a temporary absence of blood flow in the carotid artery. The duration of this period is a crucial characteristic of this type of surgery. The absence of blood flow leads to brain ischemia which is the risk factor of postoperative neurocognitive disorders such as emergence delirium, postoperative delirium and postoperative cognitive dysfunction.

Some surgical and non-surgical methods for brain protection were evaluated. According to recent data, there is no evidence of effective pharmacological protective methods that can decrease brain damage during carotid artery surgery.

Nevertheless, some trials demonstrated that using lithium-based medications for patients with a stroke can reduce the volume of the stroke. Therefore, the investigators want to check the hypothesis that using lithium-based medication in the preoperative period can reduce brain damage during carotid artery surgery.

The objectives of this trial:

To determine if Lithium carbonate is superior to placebo for the occurrence of emergence delirium, agitation, postoperative delirium and postoperative cognitive dysfunction.

To determine if Lithium carbonate is non-inferior to placebo for the occurrence of a new arrhythmia, leukocytosis, acute kidney injury, seizure disorders, diarrhea, nausea, and vomit.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* elective carotid artery surgery
* general anesthesia
* written informed consent

Exclusion Criteria:

* urgent surgery
* recent ( < 1 month) overt stroke
* Mini-mental State Examination < 20 points
* The presence of any mental disorder according to the International Classification of Diseases 11th Revision which is confirmed by a psychiatrist.
* The presence of any neuromuscular disease according to the International Classification of Diseases 11th Revision
* Hypersensitivity or known allergy to lithium carbonate
* History of seizure disorder
* History of leukemia
* Estimated glomerular filtration rate < 30 ml/min/1.73 m2
* Left ventricular ejection fraction < 30%
* Heart failure equal 3 or 4 class according to the New York Heart Association Functional Classification
* Pregnant or breast-feeding women
* Inability to undergo a preoperative assessment for any reason
* Previously enrolled in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2021-11-20 (Actual); Primary Completion 2025-05-19 (Actual); Study Completion 2025-05-19 (Actual)

PRIMARY OUTCOMES:
Frequency of emergence delirium | 30 days
  Number of patients with positive the confusion assessment method for the intensive care unit as soon as they reach Aldrete score of 9 points

SECONDARY OUTCOMES:
Frequency of agitation | 30 days
  Richmond agitation-sedation scale more or equal +2 evaluated from the end of volatile anesthetic supply to the moment when a patient reaches Aldrete score of 9 points
  Richmond agitation-sedation scale:
  minimum value = -5 (Unarousable - no response to voice or physical stimulation) maximum value = +4 (Combative - overtly combative or violent; immediate danger to staff) Adequate patients have the results of Richmond agitation-sedation score equal 0 (Alert and calm; Spontaneously pays attention to caregiver)
Frequency of postoperative delirium | 30 days
  Number of patients with even one positive confusion assessment method for the intensive care unit or 3-minute confusion assessment method
Length of postoperative delirium | until 1 month after surgery
  30 days - number of days in which patient had positive confusion assessment method for the intensive care unit or 3-minute confusion assessment method
Frequency of overt strokes | 1 year
  Number of overt strokes
Frequency of covert strokes | 1 year
  Number of covert strokes
Length of stay in intensive care unit | 1 month
  Number of days in intensive care unit
Length of hospitalization | 1 month
  Number of days in hospital
Frequency of cardiac death | 1 year
  Number of of cardiac deaths
Frequency of non-fatal cardiac arrest | 1 year
  Number of non-fatal cardiac arrests
Frequency of major adverse cardiac event | 1 year
  Number of major adverse cardiac events
Frequency of major adverse cardiac and cognitive event | 1 year
  Number of major adverse cardiac and cognitive events
30-days mortality | 30 days
  Number of deaths in period of 30 days after surgery
1-year mortality | 1 year
  Number of deaths in period of 1 year after surgery
Frequency of new postoperative arrhythmia | 1 month
  Number of new postoperative arrhythmias
Frequency of leukocytosis | From 2 days before surgery to the day of surgery
  Number of patients with leukocytosis
Frequency of acute diarrhea | From 2 days before surgery to the day of surgery
  Number of patients with acute diarrhea
Frequency of postoperative nausea and vomit | 1 month
  Number of patients with postoperative nausea and vomit
Frequency of preoperative nausea and vomit | From 2 days before surgery to the day of surgery
  Number of patients with preoperative nausea and vomit
Frequency of acute kidney injury | 1 month
  Number of patients with acute kidney injury
Frequency of myasthenia | From 2 days before surgery to the day of surgery
  Number of patients with myasthenia
Frequency of preoperative seizure | From 2 days before surgery to the day of surgery
  Number of patients with seizure
Frequency of postoperative seizure | 1 month
  Number of patients with seizure
Serum level of S100 beta protein | 2 days after surgery
  Serum level of S100 beta protein
Serum level of neuron-specific enolase | 2 days after surgery
  Serum level of neuron-specific enolase
Serum level of Tau-protein | 2 days after surgery
  Serum level of Tau-protein
Serum level of Neurofilament light polypeptide | 2 days after surgery
  Serum level of Neurofilament light polypeptide
Serum level of Glial fibrillary acidic protein | 2 days after surgery
  Serum level of Glial fibrillary acidic protein

CONTACTS AND LOCATIONS:
Overall Officials: Valery Likhvantsev, PhD, Principal Investigator — Negovsky Reanimatology Research Institute
Locations (1):
- Demikhov Municipal Clinical Hospital 68, Moscow, Russia